CLINICAL TRIAL: NCT03147768
Title: Phase I Feasibility Trial To Study The Safety Of Sealing Resected Pancreatic Surfaces After Partial Distal Pancreatectomy Using Laser Tissue Welding
Brief Title: Laser Tissue Welding - Distal Pancreatectomy Sealing Study
Acronym: LTW
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laser Tissue Welding, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); CHI St. Luke's Health, Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Phase I - LTW Pancreas Sealing; R44CA203052 (NIH)
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Tumor, Benign; Pancreatic Neoplasms; Pancreatic Adenocarcinoma; Pancreatic Pseudocyst; Pancreatic Neuroendocrine Tumor; Pancreas; Insulinoma; Pancreatic Cyst; Pancreatic Teratoma; Pancreatic Polypeptide Tumor; Pancreatic Vipoma; Pancreatic Cystadenoma; Pancreas Injury; Pancreatic Gastrinoma; Pancreatic Glucagonoma
Keywords: Laser Tissue Welding; Pancreatic Sealing; Hemostasis; Pancreatic Tumors; Pancreatic Resection; Pancreatic leakage; LTW
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Pseudocyst; Adenoma, Islet Cell; Insulinoma; Pancreatic Cyst; Vipoma; Glucagonoma

STUDY DESIGN:
Intervention Model Description: Open Label Combination Product (Laser + Biologic + Drug) regulated as a device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Distal Pancreatectomy Sealing using LTW (Experimental): At the completion of pancreatic resection, the cut surface of the pancreas is covered with two layers of Albu-Green solder and one layer of D-Albumin lamina, all welded with the laser. The 60 Watt custom 810nm diode laser, is set to deliver continuous energy with laser irradiation power of approximately 150 W/cm2 with a Fluence of 90 J/cm2. During soldering the tip of the custom hand piece with top hat beam profile is held 1-2 cm from the wound surface to generate a 5mm spot size. Albu-Green Solder is observed to convert from a liquid green state to a solid white crust when the laser is activated indicating the completion of welding and providing a visual cue to the operator. The amount of Albu-Green solder and size of the denatured albumin lamina used is documented. The total laser tissue welding time for the three layers and the laser tissue welding time in seconds per cm2 is documented.
  Interventions: Device: Distal Pancreatectomy Sealing Using LTW

INTERVENTIONS:
Device: Distal Pancreatectomy Sealing Using LTW — The device's intended use is to seal the pancreatic surface using a laser to weld human albumin based biomaterials after surgical removal of pancreatic tumors during a partial pancreatectomy.

SUMMARY:
The laser tissue welding device is intended for use in patients requiring sealing of the pancreas after partial pancreatectomy, and including those patients who are fully heparinized or have hemodilutional coagulation failure.

The hypothesis is that the laser tissue welding device is safe and effective in sealing the pancreas, thereby decreasing the blood loss (operative and post-operative), and pancreatic juice leakage for patients when the Laser Tissue Welding device is used after pancreatic resection.

DETAILED DESCRIPTION:
UNMET CLINICAL NEED

In the United States, pancreatic cancer is the fourth leading cause of cancer-related death in both men and women and will be the second leading case by 2030. Pancreatoduodenectomy (Whipple procedure) and distal partial pancreatectomy is used to treat pancreatic tumors, and these procedures are associated with a high rate of morbidity due to pancreatic fistulae.

As per the Surveillance, Epidemiology and End Results (SEER) Program: It is estimated that 41,609 men and women (21,370 men and 21,770 women) will be diagnosed with and 38,460 men and women will die of cancer of the pancreas in 2013. The five-year survival is dismal, 24.1% for localized malignancy, and drops to 6% if there is regional spread. There are 45,220 new cases in 2013 and 38,460 deaths.

Distal Pancreatectomy may be indicated for malignant exocrine tumors of the body and tail of pancreas (62%), insulinomas, chronic pancreatitis (12%), pancreatic pseudocysts, non pancreatic tumors (23%) and injury due to trauma.

Due to heighten awareness and preventative care, there has been an increase in detection of incidental small pancreatic mass cases due to widespread use of abdominal cross sectional imaging and thus an increase in the amount of pancreatic surgery performed. This is the stage when curative resections may be possible.

1. Surgical removal of the tumor is the only chance of a cure at T1A.
2. All pancreatic tumors at any stage require bulk reduction by a surgical procedure.

For patients undergoing distal pancreatectomy, pancreatic fistulas occurred post-operatively in 31% of patients. Over the long-term Kazanjian et al analyzed, 182 patients from 1996-2005 who underwent Pancreatoduodenectomy to treat ductal adenocarcinoma, concluded that the principal factor influencing long-term survival was operative blood loss. Pancreatic fistula is a main cause of postoperative morbidity, and is associated with numerous further complications, such as intra-abdominal abscesses, wound infection, sepsis, electrolyte imbalance, malabsorption, and hemorrhage, and with a dramatically increase in healthcare resource utilization.

The current state-of-art pancreatic surgical resections have an unacceptable pancreatic leak rate of 30-50%. This is because there are no FDA cleared or approved sealants or devices found to be safe or effective for sealing this organ. The current standard of care is anything but standard because of the use of off-label devices and sealants.

* Endo GIA Staplers: 510 (k) k111825 Cleared on basis of "literature review" without animal or human safety or efficacy data.
* Gore SeamGuard staple/suture reinforcement material 510 (k) k043056 Synthetic bio absorbable glycolide and trimethylene carbonate copolymer. Cleared on basis of in-vivo studies done "without performance standards" under section 514.
* Surgical Sealants: All used "off label": None are FDA cleared or approved for pancreatic surgery. These are Floseal, TachoSil, Tisseel, BioGlue, and CoSeal.

Jörg Kleeff et al reviewed the factors for surgical failure of distal pancreatectomy in 302 consecutive patients from 1993 to 2006 using four different surgical closures (gut anastomosis, seromuscular patch, suture and stapling device). Although distal pancreatectomy is less moribund as compared to Whipple procedure, morbidity was 32-52%, pancreatic fistulas occurred in 20-33% and mortality in 2% of cases. Pancreatic fistulas contributed significantly to morbidity, sepsis, length of stay and overall costs. Stapler closure of the pancreatic remnant is associated with a significantly higher fistula rate.

Laser Tissue Welding is the first combination (laser and biologic) class III surgical device intended to join and seal tissues accurately and instantly. The treatment process uses thermal energy created when a laser excites photosensitive dye molecules, to coagulate the protein albumin which transforms from a liquid to a solid instantly. Laser tissue welding creates a non-compressive, non-ablative sealing of tissues with microscopic thermal damage. This combination of a laser with albumin biologics stops bleeding and fluid leaks in nanoseconds without using sutures, hemostatic clotting factors (platelets/thrombin/fibrin), thermal or cryoablation.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be 18 years and older of both genders.

1. T1a (≤ 4 cm, as measured by the maximal dimension by CT or MRI). Final determination of disease stage is made during the operation by the investigator. All resectable cystic, benign, primary or secondary malignant tumors.
2. Serum creatinine: ≤ 2.5 mg/dL
3. Glomerular filtration rate greater than ≥ 50 ml/min/m2
4. Platelet count ≥ 50,000/mm3
5. Prothrombin time < 18 seconds
6. PTT not >1.5 times control (except for therapeutically; anticoagulated nonrelated medical conditions [e.g., atrial fibrillation]);
7. Serum albumin levels > 3g/dL (Normal range 3.5 to 5 g/dL)

Exclusion Criteria:

1. Age younger than 18 years' old
2. Severe uncorrected hypertension (> 180 systolic and >110 diastolic)
3. Uncorrectable coagulopathies (on Plavix, Aspirin or Lovanox)
4. Pregnancy
5. Females who are breast feeding who do not switch the infant to formula prior to surgery
6. Active urinary tract infection
7. T1b (>4 cm) lesion and above
8. Systemic or local infection.
9. Subject has known allergy or intolerance to iodine or human serum albumin.
10. Recent febrile illness that precludes or delays participation preoperatively.
11. Treatment with another investigational drug or other intervention during the study and follow-up period.
12. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
PRIMARY EFFICACY AS A SEALANT: Intra-operative blood loss | Intra-operative
  Operative blood loss is defined by: volume of blood in the suction bottles, volume of blood clots, and weight of surgical towels before and after use. Clinical drop in hemoglobin (1 gm% = 300 ml) without hemodilution.
  Correlates with intra-operative blood transfusions. Correlates with post-operative blood transfusions.

SECONDARY OUTCOMES:
SECONDARY SAFETY: Post-operative blood loss requiring return to the operating room | 30 days
  Secondary hemorrhage or intra-abdominal hematoma requiring surgical evacuation
SECONDARY SAFETY: Prolonged post-operative pancreatic leakage | 30 days
  Pancreatic juice leakage is measured in drainage bottles (ml/day) following surgery till a drain placed during the operation is removed before patient discharge. Accumulation of fluids around the pancreas will be assessed with U/S and CT scan at the mentioned time points.
SECONDARY SAFETY: Surgical space abscess | 30 days
  Secondary infection, intra-abdominal abscess formation requiring surgical evacuation

OTHER OUTCOMES:
SECONDARY EFFICACY: Total operating time (minutes) | Intra-operative assessment
  Duration and Cost Metric
SECONDARY EFFICACY: Pancreas clamp time (minutes) | Intra-operative assessment
  Duration Metric: Assesses organ ischemia and handling, and will correlate with compromised function (rise in serum Amylase and Lipase) (assesses organ ischemia and will correlate with compromised function)
SECONDARY EFFICACY: Laser tissue welding time or time to hemostasis (Duration Metric) | Intra-operative assessment
  Duration and Cost Metric
SECONDARY EFFICACY: Length of ICU stays (Duration and cost Metric ) | 30 days
  Duration and Cost Metric
SECONDARY EFFICACY: Total hospital stay (Duration and cost Metric ) | 3 months
  Duration and Cost Metric

CONTACTS AND LOCATIONS:
Overall Officials: OMAR BARAKAT, M.D, Principal Investigator — Baylor CHI St. Luke's Medical Center, Houston, Texas; STEPHEN HAROLD, M.D.; MPH; CCRC, Study Director — Baylor CHI St. Luke's Medical Center, Houston, Texas
Locations (1):
- Baylor CHI St. Luke's Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleeff J, Diener MK, Z'graggen K, Hinz U, Wagner M, Bachmann J, Zehetner J, Muller MW, Friess H, Buchler MW. Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2007 Apr;245(4):573-82. doi: 10.1097/01.sla.0000251438.43135.fb. PMID 17414606
- [Background] Goh BK. Re: Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2008 Feb;247(2):392-3; author reply 393. doi: 10.1097/SLA.0b013e318164022d. No abstract available. PMID 18216551
- [Background] Kazanjian KK, Hines OJ, Duffy JP, Yoon DY, Cortina G, Reber HA. Improved survival following pancreaticoduodenectomy to treat adenocarcinoma of the pancreas: the influence of operative blood loss. Arch Surg. 2008 Dec;143(12):1166-71. doi: 10.1001/archsurg.143.12.1166. PMID 19075167
- [Background] Shrikhande SV, D'Souza MA. Pancreatic fistula after pancreatectomy: evolving definitions, preventive strategies and modern management. World J Gastroenterol. 2008 Oct 14;14(38):5789-96. doi: 10.3748/wjg.14.5789. PMID 18855976
- See also: NCI SEERS Register Cancer Stat Facts: Pancreas Cancer — https://seer.cancer.gov/statfacts/html/pancreas.html
- See also: NCI: A Snapshot of Pancreatic Cancer - Incidence and Mortality — https://www.cancer.gov/research/progress/snapshots/pancreatic
- See also: Endo GIA Staplers: 510 (k) k111825 — http://www.accessdata.fda.gov/cdrh_docs/pdf11/K111825.pdf
- See also: Gore SeamGuard staple/suture reinforcement material 510 (k) k043056 — http://www.accessdata.fda.gov/cdrh_docs/pdf4/K043056.pdf